CLINICAL TRIAL: NCT05402982
Title: Intraoperative Fluid Management of Large Volume Liposuction Surgery , Cardiometry Guided Stroke Volume Variation Versus Rohrich Formula
Brief Title: Intraoperative Fluid Management of Liposuction , Cardiometry Versus Rohrich Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Abdel Wahed Ali (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Ahmed Abdel Wahed Ali, Principal Investigator, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fluid status of liposuction
Record Dates: First submitted 2022-05-20; First posted 2022-06-02 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Lipodystrophy
Keywords: Lipodystrophy
MeSH Terms: conditions — Lipodystrophy

STUDY DESIGN:
Intervention Model Description: The study will done on 50 patients divided equally into two groups. Group A Fluid administration in the form of lactated ringer will be managed by Rohrich formula and the intraoperative fluid ratio (subcutaneous infiltration fluid plus intravenous fluid divided by total aspirate volume) will be 1.2(10). Rohrich formula represents fluid maintinance,deficit and replacement fluid ( 0.25 ml crystalloid given for each 1 ml above 4 litre of lipoaspirate).
  Group B Patients will receive fluid maintenance of lactated ringer 2 ml/kg/h, cardiometry guided SVV will be measured before and after induction then every 30 min ,it ranges between 5-15%, fluid bolus of lactated ringer 4 ml /kg over 15 min will be administered if SVV ˃ 15% .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A (Other): Fluid administration in the form of lactated ringer will be managed by Rohrich formula and the intraoperative fluid ratio (subcutaneous infiltration fluid plus intravenous fluid divided by total aspirate volume) will be 1.2(10). Rohrich formula represents fluid maintinance,deficit and replacement fluid ( 0.25 ml crystalloid given for each 1 ml above 4 litre of lipoaspirate).
  Interventions: Other: Rohrich formula
- GROUP B (Other): Patients will receive fluid maintenance of lactated ringer 2 ml/kg/h, cardiometry guided SVV will be measured before and after induction then every 30 min ,it ranges between 5-15%, fluid bolus of lactated ringer 4 ml /kg over 15 min will be administered if SVV ˃ 15% .
  Interventions: Device: Electrical Cardiometry (EC) ICON

INTERVENTIONS:
Device: Electrical Cardiometry (EC) ICON — Electrical Cardiometry (EC) ICON (Osypka Medical, Berlin, Germany) is an FDA approved device used for non-invasive measurement of some hemodynamic parameters as cardiac output,cardiac index, stroke volume,stroke volume variation, systemic vascular resistance, thoracic fluid content, ICON (index of contractility), variation of ICON,corrected flow time and systolic time ratio.The set data of EC are the height, weight,hemoglobin, Oxygen saturation(SPO2),age, gender ,blood pressure and heart rate(HR) of the patient
  Arms: GROUP B
Other: Rohrich formula — Rohrich formula and the intraoperative fluid ratio (subcutaneous infiltration fluid plus intravenous fluid divided by total aspirate volume) will be 1.2
  Arms: GROUP A

SUMMARY:
The aim of the study is to compare the hemodynamic parameters of fluid resuscitation using Rohrich formula to cardiometry guided stroke volume variation in patients undergoing large volume liposuction surgery .

DETAILED DESCRIPTION:
The study will done on 50 patients divided equally into two groups. Group A Fluid administration in the form of lactated ringer will be managed by Rohrich formula and the intraoperative fluid ratio (subcutaneous infiltration fluid plus intravenous fluid divided by total aspirate volume) will be 1.2. Rohrich formula represents fluid maintenance,deficit and replacement fluid ( 0.25 ml crystalloid given for each 1 ml above 4 litre of lipoaspirate).

Group B Patients will receive fluid maintenance of lactated ringer 2 ml/kg/h, cardiometry guided stroke volume variation will be measured before and after induction then every 30 min ,it ranges between 5-15%, fluid bolus of lactated ringer 4 ml /kg over 15 min will be administered if stroke volume variation ˃ 15% .

Electrical cardiometry will be connected to the patient before induction,the skin will be clean and dry before placing the electrodes. Four electrodes will be applied, first one is at the upper part of the anterior aspect of the neck, second one is 5 cm below the first electrode at lower part of the neck, third one at the lower left thorax in line with xiphoid process at the level of anterior axillary line and the fourth one is 5 cm below the third electrode at the level of anterior axillary line.Electrical cardiometry will be connected to the sensor cable and the patient data will be applied as (gender - age - height - weight - blood pressure -heart rate - hemoglobin and oxygen saturation).

Surgical Technique The wetting solution will be lactated ringer with epinephrine 1mg on 1 litre so concentration is 1:1,000,000.10 ml lidocaine 2% will be added.Subcutaneous infiltration of the wetting solution will facillate dissection and removal of fat ,the technique that will be used is traditional liposuction , suction assisted liposuction with super wet technique ( the amount of infiltration solution is equal to the amount of fat aspirate).

The liposuction cannula is a multihole blunt tip cannula with a diameter of 3 to 6 mm, 4-6 mm for deep liposuction,2-4 mm for superficial liposuction and a length ranging between 10 to 30 cm. The surgeon will inject the wetting solution to the target area until it becomes tense then infiltrates the other side waiting 10 to 15 min after infiltration to begin suction .The aspirate will be collected in suction container, fat will separate from solution after approximately 1-2 h by gravity into upper yellowish part includes fat called supernatant and lower part includes blood tinged fluid called infranatant.

Measurements

* Noninvasive blood pressure ,oxygen saturation, Heart rate before induction, 5 min and 15 min after induction then every 30 min.
* Urine output, baseline and every hour.
* Venous blood sample for measurement of hemoglobin and hematocrit level after aspiration of 4 litre of fat and for every litre after.
* Measurement of blood volume in aspirate by taking a sample from infranatant part after its separation from fat for hemoglobin level calculation and by equation of multiplying this hemoglobin concentration to infranatant volume divided by preoperative hemoglobin concentration, the investigators can measure blood volume in aspirate .
* Amount of intravenous and infiltration fluids.
* Amount of fat and total aspirate.
* Stroke volume variation before and after induction then every 30 min.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged between 21 to 60 years.
* American Society of Anesthesiologists (ASA) Ӏ& ӀӀ.
* Large volume liposuction.

Exclusion Criteria:

* Any bleeding& coagulation disorders.
* Patients on regular anticoagulant or antiplatelet drugs.
* History of previous surgery in treated areas.
* Significant cardiopulmonary, hepatic or renal disease.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-06-25 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Mean arterial blood pressure | 1 year
  Mean arterial blood pressure at 4 litre aspiration of fat and at every litre aspirated after.

SECONDARY OUTCOMES:
blood loss | 1 year
  estimation of blood loss by venous sample and suction sample
urine output | 1 year
  detection of tissue perfusion by urine output every hour

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Abdel Wahed Ali, physician, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

REFERENCES:
- [Background] Rajput RS, Das S, Chauhan S, Bisoi A, Vasdev S. Comparison of cardiac output measurement by noninvasive method with electrical cardiometry and invasive method with thermodilution technique in patients undergoing coronary artery bypass grafting. World Journal of Cardiovascular Surgery. 2014;2014
- [Background] Rohrich RJ, Leedy JE, Swamy R, Brown SA, Coleman J. Fluid resuscitation in liposuction: a retrospective review of 89 consecutive patients. Plast Reconstr Surg. 2006 Feb;117(2):431-5. doi: 10.1097/01.prs.0000201477.30002.ce. PMID 16462322
- [Background] Kadafi KT, Latief A, Pudjiadi AH. Determining pediatric fluid responsiveness by stroke volume variation analysis using ICON(R) electrical cardiometry and ultrasonic cardiac output monitor: A cross-sectional study. Int J Crit Illn Inj Sci. 2020 Jul-Sep;10(3):123-128. doi: 10.4103/IJCIIS.IJCIIS_87_18. Epub 2020 Sep 22. PMID 33409126